CLINICAL TRIAL: NCT06810700
Title: The Association Between Time in Range With Markers of Endothelail an Dcardiovascular Function in Patients With type1 Diabetes Mellitus and Minimed 780G
Brief Title: The Association Between Time in Range With Markers of Endothelial and Cardiovascular Function
Status: Not yet recruiting | Type: Observational
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, VAIA LAMBADIARI, Professor of Internal Medicine-Endocrinology, Attikon Hospital
Other Study IDs: TYPE 1DM_Time in range
Record Dates: First submitted 2025-01-31; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Type 1 Diabetes Mellitus: In this observaltional study, 90 patients aged >12 years old with T1DM who are on MiniMed 780G system will be included.We aim to investigate the association between markers of endothelial and cardiovascular function with with CGM and insulin metrics, as well as anthropometric measurements, BM, lipid levels, blood pressure.
  Interventions: Device: MiniMed 780G

INTERVENTIONS:
Device: MiniMed 780G — patients aged >12 years old with T1DM who are on MiniMed 780G

SUMMARY:
In this observaltional study, 90 patients aged >12 years old with T1DM who are on MiniMed 780G system will be included.We aim to investigate the association between time in range (70-140mg/dl) and time in tight range (70-180mg/dl) with markers of endothelial and cardiovascular function.

DETAILED DESCRIPTION:
In this observational study, 90 participants with T1D on MiniMed 780G system will be included. HbA1c, anthropometric measurements, CGM and Insulin Metrics will be assessed in all patients. Moreover, the investigators will assess:

1. the pulse wave velocity, the augmentation index and the central systolic blood pressure which are markers of arterial stiffness
2. the perfused boundary region of subglingulal vessels which is marker of endothelial function
3. the global longitudinal strain which is marker of myocardial function.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 1 diabetes >1 year prior to consent date. Diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not required.
2. HbA1c < 12.5%
3. Age >7years at the initiation of the system
4. Multiple Daily Injections (Basal Bolus therapy) with Total daily insulin use of great than 8.0 units per day over a 1-week period
5. Clinically able to start the AHCL system
6. History of 3 clinic visits in the last year

Exclusion Criteria:

1. Diabetic Ketoacidosis in the 6 months prior to screening visits

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients aged >12 years old with T1DM who are on MiniMed 780G system .
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Endothelial glycocalyx | Baseline
  The association between time in range and the thickness of endothelial glycocalyx
Pulse wave velocity | Baseline
  The association between time in range and pulse wave velocity
Global longitudinal strain | Baseline
  The association between time in range and global longitudinal strain